CLINICAL TRIAL: NCT01842880
Title: Validation of MicroRNAs as Biomarkers for Determining Patients Prognosis With Chagas Disease
Brief Title: MicroRNAs as Biomarkers in Patients With Chagas Disease
Status: Completed | Type: Observational
Sponsor: Hospital Sao Rafael (Other)
Responsible Party: Principal Investigator, Milena Botelho Pereira Soares, PhD, Hospital Sao Rafael
Other Study IDs: CEP-41-10-2
Record Dates: First submitted 2013-04-23; First posted 2013-04-30 (Estimated); Last update posted 2015-02-20 (Estimated); Status verified 2015-02

CONDITIONS: Chagas Disease
Keywords: MicroRNAs; Chagas disease; Biomarkers
MeSH Terms: conditions — Chagas Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Plasma, Serum, Whole Blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients with Chagas disease diagnosis: Diagnosis of Chagas disease in both forms: indeterminate and cardiac ones, with and without ventricular dysfunction.

SUMMARY:
The purpose of this study is to analyze the efficacy of MicroRNAs as biomarkers on the Chagas Disease prognosis. This analysis will be done through the correlation between the plasmatic levels of this molecule with functional and laboratory tests.

DETAILED DESCRIPTION:
The patients included in the study must at first sign the written consent. They shall be accompanied in the specialized outpatient clinics for Chagas disease - Hospital São Rafael - Centro de Biotecnologia e Terapia Celular. They will be submitted to several tests, including:

* Collection of Blood samples for biochemical analysis;
* Electrocardiogram;
* Holter Electrocardiogram;
* Echocardiogram;
* Treadmill Test;
* X-Ray Imaging;
* Magnetic Resonance Imaging;
* Evaluation of the quality of life through the application of questionnaires (SF 36 and the Minnesota Living With Heart Failure Questionnaire).

ELIGIBILITY:
Inclusion Criteria:

* Chagas disease diagnosis confirmed by 2 different serologies
* Diagnosis of Chagas disease in both forms: indeterminate and cardiac ones, with and without ventricular dysfunction.

Exclusion Criteria:

* Significant valve disease defined as aortic stenosis with a gradient of VE/Ao > 50 mmHg
* Mitral stenosis with a valve area inferior than 1,5 cm2
* Severe or moderate aortic and/or mitral regurgitation
* Chronic use of immunosuppressive agents
* Dialysis treatment of terminal renal failure
* Fever on the last 48 hours or evidence of systemic infection in activity according to the definition of sepsis of the ACCP/SCCM (American College os Chest Physicians/Society of Critical Care Medicine)
* Current abusive use of alcohol or illicit drugs (Based on the DSM IV)
* Any other comorbidities that impact patient's survival within the next 2 years
* Liver disease in activity
* Continuous use of steroids as treatment for COPD
* Hematologic, neoplastic or bone diseases
* Homeostasis disturbances
* Inflammatory diseases or chronic infectious diseases

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Tertiary Hospital
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2011-01; Primary Completion 2013-06 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Correlation of plasmatic levels of MicroRNAs with the percentage of heart fibrosis | One year
  Mensuration of heart fibrosis percentage with Magnetic Resonance Imaging

SECONDARY OUTCOMES:
Correlation of plasmatic levels of MicroRNAs with the functional cardiovascular capacity | One year
  Mensuration of the functional capacity with treadmill test.
Correlation of plasmatic levels of MicroRNAs with the left ventricular function | One year
  Mensuration of the left ventricular function with echocardiogram and magnetic resonance imaging
Correlation of plasmatic levels of MicroRNAs with the serum levels of Pro-BNP. | One year
Correlation of plasmatic levels of MicroRNAs with the serum levels of TNF-alpha | One year
Correlation of plasmatic levels of MicroRNAs with the serum levels of IFN-gamma. | One year

CONTACTS AND LOCATIONS:
Overall Officials: Milena Botelho Pereira Soares, PhD, Principal Investigator — Hospital São Rafael; Ricardo Ribeiro dos Santos, MD, Study Director — Hospital São Rafael; Ticiana Ferreira Larocca, MD, Study Chair — Hospital São Rafael; Márcia Maria Noya Rabelo, MD, Study Chair — Hospital São Rafael; Luís Cláudio Lemos Correia, MD, Study Chair — Hospital São Rafael; Bruno Solano de Freitas Souza, MD, Study Chair — Hospital São Rafael; Carolina Thé Macedo, MD, Study Chair — Hospital São Rafael; Ana Luiza Dias Angelo, PhD, Study Chair — Hospital São Rafael
Locations (1):
- Hospital São Rafael, Salvador, Estado de Bahia, Brazil